CLINICAL TRIAL: NCT06084676
Title: Organoid Model Predictive of Response to Immunotherapies
Status: Terminated | Type: Observational
Why Stopped: difficulty recruiting participants
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Mateusz Opyrchal, Associate Professor of Medicine, Vera Bradley Foundation Scholar in Breast Cancer, Program Leader - Phase 1, Indiana University
Other Study IDs: CTO-IUSCCC-0804
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Immunotherapy — Organoid samples will be collected at time of biopsy and cultured in the lab. The samples will then receive the same standard of care immunotherapy treatment as the patient.

SUMMARY:
The purpose of this study is to create models out of tissue samples and treat those models with the same immunotherapy treatment the patient will be receiving, in order to validate this process and to predict responses to therapies and use it to choose the best treatments for people in the future. The researchers will then examine the direct effects of the treatment on those models.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Biopsy proven diagnosis of cancer
4. Able to obtain at least 2 16 gage cores of fresh tissue safely (3 or more cores preferred)
5. Planning to undergo standard of care Immunotherapy
6. Baseline standard of care CT within 8 weeks of starting Immunotherapy

Exclusion Criteria:

1. Inability to provide fresh biopsy sample
2. Any active infections
3. Any conditions that in the opinion of treating physician and the study team will compromise the ability of the patient to receive prescribed treatment to assess the response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are planning on receiving a fresh biopsy sample will be identified in the IU Oncology outpatient clinics or by referral from outside physicians.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Calculate overall patient response rate | Baseline to 12 months
  Compare patient response using RECIST 1.1 criteria and immune-organoid response based on the following criteria:
  1. Complete response <50% of viable tumor cells
  2. Response >50%<70% of viable tumor cells
  3. Stable >70%<90% viable tumor cell left
  4. Progressive >90% of viable tumor cell left
Reliability of organoid development | Baseline to 2 months
  calculate the percentage of biopsies with successful organoid development

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Opyrchal, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States